CLINICAL TRIAL: NCT05761353
Title: Endermologie Versus Negative Pressure Therapy on Postmastectomy Lymphedema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rayda Maher Mohamed Abdelkhalek, assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/003744
Record Dates: First submitted 2023-02-13; First posted 2023-03-09 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Mastectomy; Lymphedema
MeSH Terms: conditions — Lymphedema | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (endermologie group) (Experimental): This group includes 34 patients who will receive 30 min Endermologie 3 times per week in addition to their physical therapy program (active range of motion and elevation); hygiene and skin care for 6 weeks.
  Interventions: Device: Endermologie
- Group B (Negative pressure therapy group) (Experimental): This group includes34 patients who will receive 30min negative pressure therapy 3 times per week in addition to their physical therapy program (active range of motion and elevation); hygiene and skin care for 6 weeks
  Interventions: Device: Negative pressure therapy

INTERVENTIONS:
Device: Endermologie — Group A will receive -18 sessions by Endermologie system used to decrease postmastectomy lymphedema for group (A), three sessions per week for six weeks.
  Each session was 30 minutes at the posterior thorax, upper arm, forearm and the hand.
  -In addition to physical therapy program (active range of motion and elevation); hygiene and skin care
  Arms: Group A (endermologie group)
Device: Negative pressure therapy — Group B will receive negative pressure therapy with
  * Pressure: 20-250 mmHg.
  * Total treatment period: 6weeks
  * A number of sessions: 3sessions/ week. Time of application : 30 min
  * In addition to physical therapy program (active range of motion and elevation); hygiene and skin care
  Arms: Group B (Negative pressure therapy group)

SUMMARY:
Statement of the problem:

The problem will be stated in a questionary form:

"Which will be more effective endermologie or negative pressure therapy in reducing limb circumference and volume in postmastectomy lymphedema?".

Hypothesis:

It will be hypothesized that:

There is no significant difference between endermologie and negative pressure therapy in reducing circumference and limb volume in post mastectomy lymphedema.

DETAILED DESCRIPTION:
Subject:

Sixty- eight women treated for unilateral breast cancer with secondary upper limb lymphedema post mastectomy will participate in this study. Their ages will be ranged from 40 to 60 years, they will be free from any other diseases that will affect or influence the results and the participants will be selected from National Cancer Institute and randomly distributed into two equal groups in number.

Study design:

In this study the patients will be randomly assigned into two groups equal in number (34 patients for each group).

Inclusion Criteria:

The subject selection will be according to the following criteria:

* Only females will participate in the study.
* Patients' age will be ranged between 40-60 years.
* All patients will suffer from post mastectomy lymph-edema.
* All patients have a modified radical mastectomy.
* All patients will suffer from grade II lymph edema without skin changes one year post mastectomy.
* All patients are right-dominant hand.
* All patients enrolled to the study have their informed consent.

Exclusion Criteria:

The potential participants will be excluded if they meet one of the following criteria:

* primary lymph-edema.
* Diabetes mellitus.
* Pregnancy.
* Recurrent cancer.
* Current or recent cellulitis.
* Current metastases.
* Venous thrombosis.
* Photosensitivity.
* Phlebitis in development stage.
* Infection.
* Receiving anti-coagulant treatment.

Equipment:

The study equipment's will be divided into measurement and therapeutic equipment and tools:

1: Measurement equipment

1(a):Limb volume measurement:

This will be performed by measuring the circumference of each segment of the limb between two consecutive circumferences as a truncated zone. The volume of the segment was calculated as:

V=h (c12+c1c2+c22 )/12π, where V is the volume of the segment, c1 and c2 are the circumferences at the ends of the segment, and h is the distance between them.

Measurement of limb volume measurement will be conducted pre-treatment and after treatment course (6 weeks).

1. (b): Measuring Disability of the arm, shoulder and hand by: .Quick DASH questionnaire (Disability of the arm, shoulder, and hand).

   * The Quick- DASH has five response options for each item from 0=no difficulty to perform or no symptoms to 5=unable to do.
   * Quick DASH scale will be conducted pre-treatment and after treatment course (6 weeks).
2. Therapeutic equipment :

2. a. Endermologie: endermologie therapy will be three sessions per week for six weeks (total 18 sessions).

The study group will receive 18 sessions by Endermologie system ( used to decrease postmastectomy lymphedema for group (A), three sessions per week for six weeks.

Each session was 30 minutes at the posterior thorax, upper arm, forearm and the hand.

2.b. Negative pressure therapy:

* Pressure: 20-250 mm Hg.
* Total treatment period: six weeks.
* A number of sessions: 3 sessions/ week. Time of application : 30 min

ELIGIBILITY:
Inclusion Criteria:

* Only females will participate in the study.
* Patients' age was ranged between 40-60 years.
* All patients will suffer from post mastectomy lymphedema.
* All patients have a modified radical mastectomy.
* All patients suffer from grade II lymphedema without skin changes one year post mastectomy(as defined by the International Society of Lymphology).
* All patients are right-dominant hand.
* All patients enrolled to the study will have their informed consent.

Exclusion Criteria:

* The potential participants will be excluded if they meet one of the following criteria:

  * primary lymphedema.
  * Diabetes mellitus.
  * Pregnancy.
  * Recurrent cancer.
  * Current or recent cellulitis.
  * Current metastases.
  * Venous thrombosis.
  * Photosensitivity.
  * Phlebitis in development stage.
  * Infection.
  * Receiving anti-coagulant treatment.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2022-06-29 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Measuring Disability of the arm, shoulder and hand | Measuring will be taken before treatment and after 6 weeks of treatment to monitor the change in upper limb function before and after treatment
  Measuring Disability of the arm, shoulder and hand will be carried out by using Quick-DASH questionnaire
Limb volume measurement | Measuring will be taken before treatment and after 6 weeks of treatment to monitor the change in upper limb volume and decrease of lymph-edema
  Limb volume measurement will be carried out by by measuring the circumference of each segment of the limb between two consecutive circumferences as a truncated zone. The volume of the segment was calculated as:
  V=h (c1+c1c2+c2 )/12π

CONTACTS AND LOCATIONS:
Overall Officials: Rayda M Mohamed, Principal Investigator — Cairo Unversity
Locations (1):
- Outpatient clinic, Faculty of Physical Therapy, Cairo university, Giza, Dokki, Egypt

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-05-17): https://cdn.clinicaltrials.gov/large-docs/53/NCT05761353/SAP_000.pdf